CLINICAL TRIAL: NCT05139914
Title: Assessment of Dapagliflozin on Vascular Health in Patients With Type 2 Diabetes
Acronym: SFRNDM2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was halted early because of the inability to enroll participants.
Sponsor: Boston University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-41648; 20SFRN35120118 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2021-11-19; First posted 2021-12-01 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; Endothelial Dysfunction
Keywords: Sodium-Glucose Cotransporter-2 (SGLT2) inhibitor; Dapagliflozin; Endothelial cell (EC) Health; Vascular function; EC gene expression levels; Circulating miRNA; Biomarkers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dapagliflozin then Placebo (Experimental): Participants in this arm will receive dapagliflozin and then placebo with a 2 week wash out period in between.
  Interventions: Drug: Dapagliflozin; Other: Placebo
- Placebo then dapagliflozin (Placebo Comparator): Participants in this arm will receive placebo and then dapagliflozin with a 2 week wash out period in between.
  Interventions: Drug: Dapagliflozin; Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg/day (in capsule form) of dapagliflozin for 6 weeks
  Other Names: Sodium-Glucose Cotransporter-2 (SGLT2) inhibitor
Other: Placebo — Placebo capsule for 6 weeks

SUMMARY:
Patients with Type 2 Diabetes Mellitus (T2DM) have changes in blood vessel health that can lead to a higher chance of developing heart attacks or strokes. New medications for T2DM including dapagliflozin, which is a Sodium-Glucose Cotransporter-2 inhibitor (SGLT2) inhibitor, may help protect the heart and blood vessels.

The overarching objective of this mechanistic study is to learn how a Sodium-Glucose Cotransporter-2 (SGT2) inhibitor, dapagliflozin, impacts vascular health in patients with Type 2 Diabetes Mellitus (T2DM). The investigators will compare the changes in vascular health to changes in endothelial cell (EC) phenotype including non-coding RNA (ncRNA) to develop evidence supporting the mechanism of cardiovascular benefit of SGLT2 inhibitors. This study will provide novel information regarding the mechanism of effects of novel treatments for endothelial function and vascular health in patients with T2DM to reduce cardiovascular (CV) risk. The research aims to assess the:

* effects of dapagliflozin on EC phenotype.
* impact of dapagliflozin on vasodilator function and additional measures of vascular health including arterial stiffness and circulating markers of vascular health.

DETAILED DESCRIPTION:
The study design is a two-treatment, two-period crossover, double-blind, placebo-controlled design study to investigate the effect of the SGLT2 inhibitor, dapagliflozin, on Endothelial Cell (EC) phenotype, EC RNA levels, circulating microRNA (miRNA), and biomarkers in patients with T2DM. Subjects will be randomized to treatment order in a 1:1 ratio to receive SGLT2 inhibitor (dapagliflozin) and then placebo or vice versa in a crossover design. Total study period for each study subject is 14 weeks consisting of: two treatment periods (dapagliflozin and placebo) lasting 6 weeks each (12 weeks total) and a 2 week washout period between treatment periods. Each subject undergoes a washout period of 2 weeks after completing first 6 weeks of treatment with either placebo or dapagliflozin. This is followed by crossover to the alternate treatment period of 6 weeks with dapagliflozin or placebo depending on their first treatment. Randomization will be done in block sizes of 2 or 4. Once assigned to treatment, participants will receive dapagliflozin 10 mg/day or placebo for 6 weeks.

The study was terminated due to the inability to enroll the anticipated 50 participants to test the research hypotheses (only 3 participants were randomized in almost 3 years). There were too few samples to test for endothelial cell related outcomes, miRNA, and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM for minimum of 3 months defined as fasting glucose greater than or equal to 120 mg/dL, hemoglobin A1C (HbA1C) ≥6.5%
* Body mass index (BMI) >25
* Willing to give written informed consent and able to understand, to participate in and to comply with the study requirements.

Exclusion Criteria:

* Treatment with anticoagulation
* Treatment with SGLT-2 inhibitor
* HbA1c >9.5% within the last 3 months
* Systolic blood pressure less than 120mm Hg
* History of genital mycotic infections: more than one genital mycotic infection in the past two years
* History of recurrent urinary tract infections: history of chronic cystitis and/or recurrent urinary tract infections (3 or more in the last year)
* History of allergy to SGLT-2 inhibitor
* History of bladder cancer or prior pelvic radiation
* More than one hypoglycemic events in the past 6 months and/or HbA1c <7.0%
* Women lactating or pregnant. All women with childbearing potential will undergo a blood pregnancy test at each visit to exclude pregnancy.
* Treatment with an investigational product within the last 30 days.
* Clinically evident major illness of other organ systems, including clinically evident cancer, renal failure (GFR<60 mL/min), or other conditions that in the opinion of the principal investigator make a clinical study inappropriate

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Hamburg, MD, Principal Investigator — BU School of Medicine, Cardiovascular Medicine
Locations (1):
- BU School of Medicine Evans 748, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 participants were enrolled but 1 was ineligible after screening so that 3 were randomized.
Period: Overall Study
Arm/Group | Dapagliflozin Then Placebo | Placebo Then Dapagliflozin
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin Then Placebo | Placebo Then Dapagliflozin | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Systolic Blood Pressure
Description: Supine blood pressures were measure in triplicate after 10 minute rest period using Omron blood pressure cuff
Time Frame: 14 weeks
Population: Data were not analyzed for either study arm as there was only one participant in each arm at 14 weeks.
Arm/Group | Dapagliflozin Then Placebo | Placebo Then Dapagliflozin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Mean Diastolic Blood Pressure
Description: Supine blood pressures were measure in triplicate after 10 minute rest period using Omron blood pressure cuff
Time Frame: 14 weeks
Population: Data were not analyzed for either study arm as there was only one participant in each arm at 14 weeks.
Arm/Group | Dapagliflozin Then Placebo | Placebo Then Dapagliflozin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Dapagliflozin Then Placebo | Placebo Then Dapagliflozin
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated due to the inability to enroll the anticipated 50 participants to test the research hypotheses (only 3 participants were randomized in almost 3 years). There were too few samples to test for endothelial cell related outcomes, miRNA, and biomarkers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT05139914/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT05139914/ICF_001.pdf